CLINICAL TRIAL: NCT06525506
Title: A Multicenter, Randomized, Double-Masked Phase II Study Evaluating the Efficacy and Safety of IBI311 in Subjects With Inactive or Active Thyroid Eye Disease
Brief Title: A Study of IBI311 in Subjects With Inactive or Active Thyroid Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI311A202
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-10

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 2: IBI311 (3-20 mg) (Active Comparator): Arm 2: IBI311 (3-20 mg). Participants will receive 8 intravenous infusions of IBI311 with an interval of 3 weeks. Dose conversion was performed at week 12.
  Interventions: Biological: IBI311 (3-20 mg)
- Arm 4: IBI311 (20 mg) (Active Comparator): Arm 4: IBI311 (20 mg). Participants will receive 8 intravenous infusions of IBI311 with an interval of 3 weeks.
  Interventions: Biological: IBI311 (20 mg)
- Arm 3: IBI311 (10 mg) (Active Comparator): Arm 3: IBI311 (10 mg). Participants will receive 8 intravenous infusions of IBI311 with an interval of 3 weeks.
  Interventions: Biological: IBI311 (10 mg)
- Arm 1: IBI311 (3-10 mg) (Active Comparator): Arm 1: IBI311 (3-10 mg). Participants will receive 8 intravenous infusions of IBI311 with an interval of 3 weeks. Dose conversion was performed at week 12.
  Interventions: Biological: IBI311 (3-10mg/kg)

INTERVENTIONS:
Biological: IBI311 (20 mg) — Arm 4: 10 mg/kg IBI311 on Day 1, followed by 20 mg/kg IBI311 from week 3 to week 21, Q3W.
  Arms: Arm 4: IBI311 (20 mg)
Biological: IBI311 (3-20 mg) — Arm 2: 3 mg/kg IBI311 from day 1 to week 9, Q3W, followed by 20 mg/kg IBI311 from week 12 to week 21, Q3W.
  Arms: Arm 2: IBI311 (3-20 mg)
Biological: IBI311 (10 mg) — Arm 3: 10 mg/kg IBI311 from day 1 to week 21, Q3W.
  Arms: Arm 3: IBI311 (10 mg)
Biological: IBI311 (3-10mg/kg) — Arm 1: 3 mg/kg IBI311 from day 1 to week 9, Q3W, followed by 10 mg/kg IBI311 from week 12 to week 21, Q3W.
  Arms: Arm 1: IBI311 (3-10 mg)

SUMMARY:
This is a multicenter, randomized, double-masked phase II study evaluating the efficacy and safety of IBI311 in subjects with inactive or active thyroid eye disease. Approximately 36 subjects meeting the study eligibility criteria will be randomly assigned to the 3-10 mg group, 3-20 mg group, 10 mg group, or 20 mg group on day 1 in a 1:1:2:2 ratio. Dose conversion of the 3-10 mg or 3-20 mg group was performed at week 12. Active and inactive TED was a stratification factor in this study. Active and inactive TED subjects were enrolled in a 1:1 ratio.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent.
2. Male or female subject between the ages of 18 and 80 years at screening.
3. Weight between 50 kg and 100 kg.
4. Moderate-to-severe active TED:

   * CAS ≥ 3 in the study eye at screening and baseline;
   * Usually associated with at least two of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement, exophthalmos ≥ 3 mm above normal, and/or inconstant or constant diplopia;
   * ≤ 12 months since the onset of active TED symptoms according to subjects' chief complaint or medical record at screening;

   Inactive TED:
   * According to subjects' chief complaint or medical record at screening, initial diagnosis of TED > 12 months but < 10 years prior to screening.
   * CAS ≤ 2 in both eyes at screening and baseline and CAS ≤ 2 in both eyes for at least 6 months prior to screening or all of the following at least 6 months prior to screening: a. no progression in proptosis; b. no progression in diplopia; c. no new inflammatory TED symptoms.
   * Exophthalmos ≥ 3 mm above normal.
5. Exophthalmos ≥ 20 mm in the study eye at baseline.
6. Female subjects should be fertile women who are sterile or have a negative blood pregnancy test during the screening period and who agree to take contraceptive measures within 120 days from the screening period to the last medication; Male subjects should agree to use contraception from the screening period to 120 days after the last dose.

Key Exclusion Criteria:

Subjects will be ineligible for study participation if they meet any of the following criteria:

1. Baseline CAS decreased by ≥ 2 points, or baseline proptosis decreased by ≥ 2 mm as compared with screening.
2. Visual function impairment due to optic neuropathy, defined as ≥ 2 lines of vision loss, new visual field defect, or color vision impairment secondary to optic nerve involvement within the past 180 days;
3. Corneal ulcers with no relief after treatment as determined by the investigator;
4. TED patients who need immediate corticosteroid therapy, orbital radiotherapy, or orbital decompression;
5. At any time prior to baseline or during the study period planned to receive orbital radiation therapy or TED surgery, including orbital decompression, strabismus surgery, and eyelid retraction correction;
6. Poorly controlled thyroid function, which was defined as free triiodothyronine (FT3) or free tetraiodothyronine (FT4) deviated more than 50% from the normal reference range of the local research center laboratory at screening.
7. Either ear had a history of tinnitus or other hearing impairment; or abnormal pure tone audiometry (defined as mean bone conduction threshold [0.5, 1, 2, 4 kHz] ≥25 dB or any bone conduction threshold ≥ 40 dB);
8. Poorly controlled diabetes at screening, defined as HbA1C ≥ 9.0% at screening, or any new medication for diabetes within 60 days prior to screening, or any dose adjustment for diabetes drugs > 10%);
9. Systemic use of glucocorticoids ≤ 30 days prior to screening;
10. Periorbital use of glucocorticoids ≤ 90 days prior to screening;
11. Systemic use of immunosuppressants ≤ 90 days prior to screening;
12. Use glucocorticoid eye drops or immunosuppressive eye drops ≤ 30 days prior to screening

12. Use IBI311 or TEPEZZA at any time prior to screening; 13 Use CD20 antibody ≤ 1 year prior to screening, or IL-6R antibody ≤ 180 days prior to screening; 14. Subjects had participated in other interventional clinical trials ≤ 90 days prior to screening, or attempting to participate in other clinical trials during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline in proptosis in the study eye. | Week 12
  Proptosis assessment: protrusion of the eye from the orbital rim as measured by Hertel exophthalmometer.
Safety and Tolerability | After receiving IBI311 treatment for 48 weeks
  Incidence, severity, and association with the study drug of ocular and systemic adverse events (AE), treatment-emergent adverse events (TEAE), and serious adverse events (SAE).

SECONDARY OUTCOMES:
The proptosis responder rate in the study eye | Week 12, 24 and 48
  Defined as percentage of subjects with a ≥ 2 mm reduction from baseline in proptosis in the study eye, without deterioration [≥ 2 mm increase] of proptosis in the non-study eye.
Mean change from Baseline in proptosis in the study eye. | Week 24 and 48
  Proptosis assessment: protrusion of the eye from the orbital rim as measured by Hertel exophthalmometer.
The overall responder rate in the study eye. | Week 12, 24 and 48
  Defined as participants with a reduction in clinical activity score (CAS) of ≥ 2 points, and a reduction in proptosis of ≥ 2 mm in the study eye, and no deterioration (increase in CAS of ≥ 2 points or increase in proptosis of ≥ 2 mm) in the non-study eye.
Percentage of subjects with a CAS of 0 or 1 in the study eye. | Week 12, 24 and 48
  According to the 7-item European Group on Graves' Ophthalmopathy (EUGOGO) amendment, CAS was used to evaluate clinical activity. For each of the following items, one point is given: spontaneous orbital pain, gaze evoked orbital pain, eyelid swelling that is considered to be due to active (inflammatory phase) Graves' ophthalmopathy (GO), eyelid erythema, conjunctival redness that is considered to be due to active (inflammatory phase) GO, chemosis, and inflammation of caruncle or plica. The sum of these points is the total score, with 0 indicating no clinical activity and 7 indicating the most severe clinical activity.
Mean change from Baseline in CAS in the study eye. | Week 12, 24 and 48
Positive responder rate to IBI311 treatment in the study eye. | Week 12, 24 and 48
  Defined as:
  1. ≥2 mm reduction of lid aperture;
  2. ≥1 point reduction in five-item CAS (excluding subjective, patient-reported spontaneous or gaze-evoked pain),
  3. ≥2 mm reduction in exophthalmos,
  4. ≥8° increase of eye muscle duction; Improvement in ≥2 features in the study eye without deterioration in the non-study eye
The impact of IBI311 on the quality of life. | Week 12, 24 and 48
  Changes in Graves' Ophthalmopathy Quality of Life (GO-QoL) questionnaire score
The diplopia responder rate | Week 12, 24 and 48
  Defined as subjects with a ≥ 1-point improvement in Gorman diplopia score.
The relapse rate after IBI311 treatment | Week 28, 36 and 48
  Defined as proptosis increased by ≥2 mm from baseline and/or CAS increased by ≥2 points from baseline with total CAS score ≥3 in either eye.
Systemic Pharmacokinetics profile of IBI311 | From Day 1 to week 24
  Descriptive statistics will be performed for concentration data, and the corresponding Pharmacokinetics parameters will be estimated if sufficient data are available.
Change from Baseline in MRI in the study eye. | Week 12, 24 and 48
  Changes in exophthalmia from baseline on MRI at week 12, 24, and 48; Changes in the volume and maximum thickness of extraocular muscle, orbital fat and lacrimal gland on MRI from baseline at week 12, 24 and 48; Changes in MRI signal of intraorbital tissue from baseline at week 12, 24 and 48.

CONTACTS AND LOCATIONS:
Locations (1):
- Innovent Biologics (Suzhou) Co. Ltd, Suzhou, Suzhou, China